CLINICAL TRIAL: NCT04312217
Title: Measuring Patient Experiences in a Children's Hospital With a Medical Clowning Intervention: A Case-Control Study
Brief Title: Medical Clowning and Patient Experiences in a Children's Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Aalto University (Other)
Responsible Party: Principal Investigator, Pekka Lahdenne, Head of Digital Services, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 164/13/03/03/2015
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Day Surgery
Keywords: patient experience; medical clowning

STUDY DESIGN:
Intervention Model Description: Children and their parents entering day surgery are pre-operatively exposed to medical clowning (N=38) or normal pre-operative care (N=32)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical clowning (Active Comparator): Preoperative medical clown exposure
  Interventions: Behavioral: Medical clowning
- Control (No Intervention): Normal preop care

INTERVENTIONS:
Behavioral: Medical clowning — Medical clowning
  Arms: Medical clowning

SUMMARY:
A case-control study is conducted in Helsinki Children's hospital. Altogether 70 children aged 4-17 years coming for a minor operative procedure including pre-operative cannula insertion will be included. Part of the patients will be exposed to medical clowning intervention and the reference group will be treated preoperatively as routinely without clowns. Emotions, anxiety levels, pain caused by the cannula insertion of the children will be monitored during the day. A survey on the emotions and expectations of the parents will be done.

DETAILED DESCRIPTION:
This study aims to measure experiences of children and their parents during day-surgery in hospital setting.

A case-control study is conducted in Helsinki Children's hospital. Altogether 70 children aged 4-17 years coming for a minor operative procedure including pre-operative cannula insertion will be included. Part of the patients will be exposed to medical clowning intervention and the reference group will be treated preoperatively as routinely without clowns. Emotions, anxiety levels, pain caused by the cannula insertion of the children will be monitored during the day. A survey on the emotions and expectations of the parents will be done.

A novel digital survey tool will be used to measure patient experiences before and after the insertion of a venous cannula needed for anaesthesia.

The research questions are as follows:

How does engagement with a medical clown during pre-operative cannulation impact on children and their parents' patient experience? How feasible is a novel data collection tool for measuring patient experience and the impact of an intervention on the patient experience of families?

ELIGIBILITY:
Inclusion Criteria:

* a patient coming for a day surgery (any) procedure in Helsinki Children's Hospital
* understands the Finnish language,
* between 4 and 17 years of age and
* the procedure includes the insertion of a venous cannula.

Exclusion Criteria:

* does not understand the Finnish language
* the child is under 4 years old or 18 years or older
* the procedure does not include the insertion of a cannula but for example mask anaesthesia

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in emotional status | Baseline and 2 hours
  Self reported emotions selected from a list of 11 emotional items. Assessment at baseline and after recovering from anesthesia.

SECONDARY OUTCOMES:
Change in anxiety status | Baseline and 2 hours
  Self reported anxiety at a scale 1-5. (1=none,..5=very much). Assessment at baseline and after recovering from anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Lahdenne, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki Children's Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karisalmi N, Maenpaa K, Kaipio J, Lahdenne P. Measuring patient experiences in a Children's hospital with a medical clowning intervention: a case-control study. BMC Health Serv Res. 2020 Apr 26;20(1):360. doi: 10.1186/s12913-020-05128-2. PMID 32336267